CLINICAL TRIAL: NCT03686566
Title: Pediatric Solid Tumor Metabolism [A Prospective, Single Center Study Exploring Solid Tumor Metabolism of Extra-cranial Tumors in the Pediatric Population]
Brief Title: Pediatric Solid Tumor Metabolism [A Prospective Study Exploring Metabolism of Solid Tumors in Pediatrics]
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Tanya Watt, Assistant Professor of Pediatrics, University of Texas Southwestern Medical Center
Other Study IDs: STU 052018-100
Record Dates: First submitted 2018-09-10; First posted 2018-09-27 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Neuroblastoma; Sarcoma; Pediatric Cancer
MeSH Terms: conditions — Neuroblastoma; Sarcoma; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 13C-glucose infusion: Tumor samples of patients who receive the optional 13C-glucose infusion will be studied using flux analysis and metabolomic profiling.
  Interventions: Drug: 13C-glucose
- No 13C-glucose infusion: Tumor samples of patients who do not choose to receive the optional 13C-glucose infusion will be studied using metabolomic profiling alone.
  Interventions: Other: No glucose infusion

INTERVENTIONS:
Drug: 13C-glucose — Includes standard pre-operation nursing care, 13C-glucose infusion and finger stick/IV glucose checks and storage of blood sample approximately every 30 minutes
  Other Names: U-C glucose
  Groups: 13C-glucose infusion
Other: No glucose infusion — Only includes standard pre-operation nursing care
  Groups: No 13C-glucose infusion

SUMMARY:
To explore metabolic phenotypes of children with extra-cranial solid tumors and compare these with their histopathological and genetic alterations to discover potential novel biomarkers and therapeutic targets to improve outcomes in children with high risk disease.

DETAILED DESCRIPTION:
The principal objective of this study is the metabolic characterization of pediatric solid tumors, with a particular focus on neuroblastoma (NBL) and fusion positive sarcoma (FPS), which will allow the detection of tumor specific metabolic alterations that can be exploited with the aim of developing novel therapeutic strategies and biomarkers.

Cellular metabolism studies provide insight, in a complementary way to genomics, into processes acting downstream from oncogenes and oncogenic fusion proteins, and such insight may point toward previously unrecognized therapeutic targets or onco-metabolites that are traceable as robust biomarkers for response. The investigator's new approach to use an in-vivo comprehensive analysis of metabolic reprograming in FPS/NBL has never been performed in childhood FPS/NBL and will complement genomics studies for these cancers. For this study, the investigators plan to obtain tumor samples at time of surgical biopsy/resection and study their metabolic signatures.

ELIGIBILITY:
Inclusion Criteria:

* Suspected malignancy
* Age ≤ 26 years and being cared for at Children's Medical Center
* Ability to undergo standard of care diagnostic procedure, including biopsy or resection of the tumor, in the OR or IR at CMC

Exclusion Criteria:

* Poorly controlled diabetes
* Any other medical condition that prevents administration of glucose

Max Age: 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children, adolescents and young adults through the age of 26 years old with a suspected malignant extra-cranial solid tumor.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Metabolic phenotypes | 2 years
  Upon collection of tumor samples, they will be processed and analyzed with mass spectrometry to learn how the tumor processes the labeled glucose by assessing enrichment of metabolites to identify the active metabolic pathways in each tumor (metabolic phenotype)
Compare the metabolic phenotype with the result of histopathological diagnosis and genetic alterations of the specific tumor | 2 years
  We will collect data and information from the patient's medical record including pathologic diagnosis and genetic testing results throughout their treatment

SECONDARY OUTCOMES:
Metabolic evolution of tumors over time | 2 years
  Compare tumor metabolism at different points in therapy (diagnosis, metastasis, recurrence) if the family consents to further studies as their child's condition progresses. Will compare high risk samples to low risk samples within a diagnosis (IE: high risk neuroblastoma vs low risk neuroblastoma)
Metabolic change due to chemotherapy | 2 years
  Compare tumor metabolism at different points in therapy (before vs after chemotherapy is given) if the family consents to further studies as their child's condition progresses. For example, tumor sample at time of neuroblastoma biopsy to resection a few months later prior to bone marrow transplantation.
Metabolic phenotypes and outcomes | 2 years
  Assess for correlations between metabolism and patient outcome if applicable

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Watt, MD, Principal Investigator — UTSW
Locations (1):
- UT Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnston K, Pachnis P, Tasdogan A, Faubert B, Zacharias LG, Vu HS, Rodgers-Augustyniak L, Johnson A, Huang F, Ricciardo S, Zhao Z, Mathews TP, Watt T, Leavey P, DeBerardinis RJ. Isotope tracing reveals glycolysis and oxidative metabolism in childhood tumors of multiple histologies. Med. 2021 Apr 9;2(4):395-410. doi: 10.1016/j.medj.2021.01.002. Epub 2021 Feb 23. PMID 33860280